CLINICAL TRIAL: NCT05566873
Title: Testing Multi-Level Remote Physical Activity Interventions in a National Sample of Older Women: The WHISH EnCore Trial
Acronym: WHISH EnCore
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Abby C King, Professor of Epidemiology and Population Health and of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 62096; R01AG071490 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Eligible individuals will be randomized to either a continuing remote educational physical activity program along with general human and planetary health information (control), or to the educational physical activity program plus a remote citizen science program aimed at physical and social environmental barriers to walking and other physical activities.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PA Education plus human and planetary health information (Active Comparator): Participants will continue to receive the remote "light touch" physical activity education program that they have been receiving for the past several years along with additional remote health education information to control for nonspecific factors (staff attention, participant time).
  Interventions: Behavioral: PA Education plus human and planetary health information
- PA Education plus Our Voice citizen science (Experimental): Participants will receive the remote "light touch" physical activity education program in combination with the remote Our Voice citizen science program aimed at identifying and addressing physical and social environmental barriers to and enablers of regular physical activity.
  Interventions: Behavioral: PA Education plus Our Voice citizen science

INTERVENTIONS:
Behavioral: PA Education plus human and planetary health information — One year of continuing person-level physical activity promotion and health-related information delivered primarily by mail, email, and through online scientific video presentations and exploration of freely available citizen science mobile applications
  Arms: PA Education plus human and planetary health information
Behavioral: PA Education plus Our Voice citizen science — One year of continuing person-level physical activity promotion and health-related information delivered primarily by mail and email, plus participatory citizen science activities involving neighborhood audits of the walking environment using a mobile app and remote group discussion and problem-solving around physical activity barriers
  Arms: PA Education plus Our Voice citizen science

SUMMARY:
While older women are disproportionately affected by chronic diseases and conditions associated with aging, including both physical and cognitive impairments, that can be alleviated or delayed by regular physical activity, few physical activity programs have been developed specifically with their needs in mind. This research aims to evaluate, in insufficiently active older women from the national WHISH pragmatic trial, the effects of a technology-driven "citizen science" approach to environmental physical activity barriers called Our Voice plus the ongoing "light-touch" remote physical activity educational program, compared to the "light-touch" remote physical activity educational program plus a control educational intervention that creates awareness around human and planetary health. This study will add important information on the benefits and trade-offs of combining these remotely delivered and practical behavioral health approaches to promote physical and cognitive health for the fast-expanding demographic group of U.S. older women.

DETAILED DESCRIPTION:
Older women are disproportionately impacted by a range of chronic diseases and conditions, such as cognitive impairments, that can be alleviated by regular physical activity (PA), including walking; yet they are the most inactive segment of the US population. This study's primary aim is to enhance the efficacy of a "light-touch", remotely delivered PA educational intervention for older women by testing the added impacts of an innovative, remotely delivered citizen science program to identify and address local environmental barriers to walking and other PA, called Our Voice (OV). The "light-touch" PA educational program (Encore) has been delivered since 2015 to >23,000 women >70 years that have been participating in the U.S.-wide Women's Health Initiative Strong and Healthy (WHISH) pragmatic PA trial. The study's hypothesis is that women receiving Encore+OV will show higher 12-month PA levels than women receiving Encore plus the control educational program. Additional questions include changes in cognitive function and sedentary behavior and exploring the relative costs of the two programs for PA change.

ELIGIBILITY:
Inclusion Criteria:

* Is insufficiently physically active based on National Guidelines;
* Can engage in moderate forms of walking in and around their neighborhoods;
* Owns and can use a smartphone;
* Willing to wear the study pedometer;
* No plans to move from the area over the 1 year study period;
* Willing to be randomized and engage in study assessments;

Exclusion Criteria:

* Not currently living in a nursing home or with a dementia diagnosis or other medical condition that would preclude moderate forms of physical activity outside the home or study participation.

Ages: 66 Years to 105 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean number of steps per day as measured by step counter | 12 months
  Participants will wear an Accusplit pedometer to record on the WHISH study website data entry tracking system their number of steps/day. Higher numbers of steps per day is considered a better outcome.

SECONDARY OUTCOMES:
Weekly walking minutes | 12 months
  Self-report using the Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire. CHAMPS is a self-report physical activity questionnaire that assesses weekly frequency and duration of various activities typically undertaken by midlife and older adults over the prior 4-week period (for example, self-reported walking for errands, for leisure, up hills, brisk walking). The measure has been shown to have good test-retest reliability (stability) and construct and concurrent validity, and has been shown to be sensitive to change in a variety of adult populations. It has seven frequency categories (from less than 1 hour a week to 9 or more hours per week). The minimum value (walking minutes) is 0 and there is no set maximum value. The national recommendation is for 150 minutes per week. Higher numbers on this measure are considered a better outcome.
Telephone Interview for Cognitive Status-modified (TICSm) | 12 months
  The 16-item (50-point) TICSm, which is the most widely used telephone cognitive assessment tools for older populations, and has been shown to have excellent validity and reliability in diverse groups of older adults. It correlates well with comprehensive neuropsychological assessments, is less constrained by ceiling effects than the Mini Mental State Examination (MMSE), and has been shown to be sensitive to change. A higher score on this measure is considered a better outcome.
Self-report Sedentary Behavior Questionnaire | 12 months
  This 7-item 1-week recall questionnaire has been shown to have good test-retest reliability and validity, and has been shown to be sensitive to change with intervention. A higher score is considered a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Abby C King, Ph.D, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Commensurate with current requirements, once the study data have undergone final data cleaning, analysis, and planned major publication, we will make the final data collected as part of the proposed research available in electronic form to experienced researchers who request them, as described below. The cleaned data set will be stored in a secure online data repository at Stanford University School of Medicine, along with a relevant "code book" of study variables. Given the multi-level, multi-method architecture of the data and the complexity it entails, we believe certain restrictions on data sharing are appropriate, e.g.: 1) no commercial use of the data and accompanying resources; 2) qualified users will include those with experience/expertise in analyzing and interpreting multi-dimensional data sources involving both qualitative and quantitative data methods. We will request that researchers submit a data request in writing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will aim to make the data and referenced resource from a publication available by the on-line publication date.
Access Criteria: See above plan description.